CLINICAL TRIAL: NCT05794750
Title: A Single-arm, Multicenter, Phase II Study Evaluating the Efficacy and Safety of Preoperative Short-course Radiotherapy Followed by Sequential Chemotherapy and AK104 for Locally Advanced Rectal Cancer
Brief Title: Assess the Efficacy of Radiotherapy and Sequential Chemotherapy and AK104 Before TME Surgery for Local CRC（AK104-IIT-13）
Acronym: AK104-IIT-13
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: JIN JING (Other)
Responsible Party: Sponsor-Investigator, JIN JING, Chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1244030031951808X0
Record Dates: First submitted 2023-02-19; First posted 2023-04-03 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: AK104; colorectal cancer; Pelvic short-course radiotherapy; TME surgery; pCR
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunotherapy; Surgical Procedures, Operative; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AK104 injection++chemotherapy (Experimental): Local CRC with short-course radiotherapy followed by sequential chemotherapy and AK104
  Interventions: Drug: AK104 injection; Procedure: TME surgery; Drug: Capecitabine; Drug: Oxaliplatin
- TME surgery (Experimental): Local CRC with short-course radiotherapy followed by sequential chemotherapy and AK104
  Interventions: Drug: AK104 injection; Procedure: TME surgery; Drug: Capecitabine; Drug: Oxaliplatin
- chemotherapy (Experimental): Local CRC with short-course radiotherapy followed by sequential chemotherapy and AK104
  Interventions: Drug: AK104 injection; Procedure: TME surgery; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: AK104 injection — Eligible subjects will receive short-course radiotherapy (SCRT), IMRT/VMAT, pelvic 25Gy/5f/1 week. Two weeks after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with immunotherapy regimen for 4 cycles: AK104 10 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W. Neoadjuvant therapy was assessed 2 weeks after the end of neoadjuvant therapy, and TME surgery was performed 4 weeks after the end of neoadjuvant therapy (R0 surgery was performed).
  Other Names: Immunotherapy
Procedure: TME surgery — Eligible subjects will receive short-course radiotherapy (SCRT), IMRT/VMAT, pelvic 25Gy/5f/1 week. Two weeks after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with immunotherapy regimen for 4 cycles: AK104 10 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W. Neoadjuvant therapy was assessed 2 weeks after the end of neoadjuvant therapy, and TME surgery was performed 4 weeks after the end of neoadjuvant therapy (R0 surgery was performed).
  Other Names: Surgery
Drug: Capecitabine — Eligible subjects will receive short-course radiotherapy (SCRT), IMRT/VMAT, pelvic 25Gy/5f/1 week. Two weeks after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with immunotherapy regimen for 4 cycles: AK104 10 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W. Neoadjuvant therapy was assessed 2 weeks after the end of neoadjuvant therapy, and TME surgery was performed 4 weeks after the end of neoadjuvant therapy (R0 surgery was performed).
  Other Names: Chemotherapy drug
Drug: Oxaliplatin — Eligible subjects will receive short-course radiotherapy (SCRT), IMRT/VMAT, pelvic 25Gy/5f/1 week. Two weeks after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with immunotherapy regimen for 4 cycles: AK104 10 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W. Neoadjuvant therapy was assessed 2 weeks after the end of neoadjuvant therapy, and TME surgery was performed 4 weeks after the end of neoadjuvant therapy (R0 surgery was performed).
  Other Names: Chemotherapy drug

SUMMARY:
This study is a single-arm, open-label, multicenter clinical study to evaluate the efficacy and safety of preoperative short-course radiotherapy combined with AK104 and chemotherapy + TME surgery in patients with advanced rectal cancer.

DETAILED DESCRIPTION:
Studies included a screening period (no more than 28 days after participants signed informed consent form to 28 days before first dose), treatment (receiving appropriate treatment until disease progression, intolerable toxicity, withdrawal of informed consent, death or study end, whichever occurs first), and follow-up (including safety follow-up and survival follow-up).

Eligible subjects will receive short-course radiotherapy (SCRT), IMRT/VMAT, pelvic 25Gy/5f/1 week. Two weeks after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with immunotherapy regimen for 4 cycles: AK104 10 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W. Neoadjuvant therapy was assessed 2 weeks after the end of neoadjuvant therapy, and TME surgery was performed 4 weeks after the end of neoadjuvant therapy (R0 surgery was performed). Patients are not recommended to enter the organ preservation observation; If the efficacy after preoperative chemoradiotherapy is evaluated as clinical complete remission (cCR) and the patient strongly refuses surgery, the patient should be informed of the risk of recurrence and ask the patient to sign a rejection of surgery. Medication safety is assessed and, depending on the severity of adverse events (AEs) and drug relevance, investigators will take steps to ensure subject safety. After surgery (or patients who strongly refuse surgery) there is a 30- and 90-day safety follow-up, and survival assessments are performed every 3 months to obtain survival information and collect new tumor treatment information until the death of the participant, withdrawal of informed consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, gender is not limited;
* 2. Stage II/III under MRI or endoscopic ultrasound ;
* 3. Fiber colonoscopy or diagnosis examination, the lower boundary of the lesion is 15m ≤ from the margin;
* 4. Rectal adenocarcinoma confirmed or revisited by pathology;
* 5. Karl Fischer score ≥ 80 points or ECOG score of 0-1;
* 6. Meet the following laboratory diagnostic indicators: hemoglobin ≥ 100g/L, white blood cell ≥ 3.5×109/L; neutrophils≥ 1.5×109/L, platelet ≥ 100×109/L; creatinine ≤ 1.0× upper limit of normal (UNL), urea nitrogen (BUN) ≤ 1.0× upper limit of normal (UNL); Alanine aminotransferase (ALT) ≤1.5× upper limit of normal (UNL); Aspartate aminotransferase (AST) ≤1.5× upper limit of normal (UNL); Alkaline phosphatase (ALP) ≤1.5× upper limit of normal (UNL); Total bilirubin (TBIL) ≤ 1.5× upper limit of normal (UNL); urine protein (-); Clotting time is normal.
* 7. No history of allergy to 5-Fu drugs, no history of allergy to platinum drugs;
* 8. With primary rectal cancer required to undergo surgery (except palliative ostomy), chemotherapy or other anti-tumor therapy before diagnosis to enrollment;
* 9. Not received radiation before;
* 10. Sign the informed consent form.

Exclusion Criteria:

* 1. Previous anti-PD-1/L1 and anti-CTLA-4 immune drugs or other immunoassay drugs;
* 2. With severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granulomatosis), etc.;
* 3. Symptomatic interstitial lung disease or active infection/non-infectious pneumonia;
* 4. Patients have risk factors for intestinal perforation: active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal cancer or other known risk factors for intestinal perforation;
* 5. History of other malignant tumors, excluding curable non-melanogenic skin cancer and carcinoma in situ of the cervix;
* 6. Active infection, heart failure, myocardial infarction, unstable angina or unstable arrhythmia within 6 months;
* 7. Physical examination or clinical laboratory findings that the investigator believes may interfere with the results or increase the patient's risk of treatment complications, or other uncontrollable diseases;
* 8. Breastfeeding or pregnant women;
* 9. Congenital or acquired immunodeficiency diseases including human immunodeficiency virus (HIV), or organ transplantation, allogeneic stem cell transplantation;
* 10. Known active hepatitis B virus (HBV), hepatitis C virus (HCV), active tuberculosis infection;
* 11. Vaccinated against tumors, or received other vaccines within 4 weeks before starting treatment (Note: Because the seasonal influenza vaccine for injection is mostly an inactivated vaccine, it is allowed to be vaccinated, while intranasal preparations are usually live attenuated vaccines, so it is not allowed)
* 12. Use other immunological agents, chemotherapy drugs, drugs in other clinical studies, and long-term cortisol therapy are not enrolled
* 13. With mental illness, substance abuse, and social problems that affect compliance will not be enrolled after a doctor's review
* 14. Allergic or contraindicated to the treatment of drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-24 (Estimated); Primary Completion 2027-04-24 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) | From date of randomization until the date of end of treatment,about 18 weeks.
  To assess the result from pathology report

SECONDARY OUTCOMES:
Major pathologic response rate (MPR) | From date of randomization until the date of end of treatment,about 18 weeks.
  To assess the result from pathology report
3-years DFS rate | From date of randomization until the date of first documented disease relapse or date of death from any cause, whichever came first about 3years..
  To compute the length between end of treatment and relapse
3-years OS rate | From date of randomization until date of death from any cause,about 3 years.
  To compute the length between end of treatment and death
Incidence and severity of adverse events (AEs) and clinically meaningful abnormal laboratory test results | From date of randomization until the date of end of treatment,about 18 weeks.
  To assess the result from inspection paper during the trail

OTHER OUTCOMES:
Relationship between the expression of immune markers in tumor tissues and blood,the distribution of immune cells, and the efficacy and prognosis of patients | From date of randomization until the date of end of treatment,about 18 weeks.
  To use PCR to check the immune markers in blood and use immunofluorescent cytochemical techniques to check the immune markers in tumor tissues.The concentration of antigens and antibodies in the blood is measured to determine the efficacy and concentration of the drug after the subject's medication

REFERENCES:
- [Derived] Xu T, Feng L, Zhang W, Li H, Ma H, Abulimiti M, Tan Y, Deng F, Huang W, Zou S, Kang W, Jiang L, Wang Y, Hu C, Chen Y, Zhou H, Tang Y, Jin J. The efficacy and safety of short-course radiotherapy followed by sequential chemotherapy and Cadonilimab for locally advanced rectal cancer: a protocol of a phase II study. BMC Cancer. 2024 Apr 19;24(1):501. doi: 10.1186/s12885-024-12254-1. PMID 38641773